CLINICAL TRIAL: NCT03830086
Title: Regional Anesthesia Versus General Anesthesia in Patients Undergoing Laparoscopic Gynecological Surgery
Brief Title: Regional Anesthesia Versus General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Mohamed Mabrouk, Principal Investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 160/2016/O/Oss
Record Dates: First submitted 2019-01-12; First posted 2019-02-05 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Postoperative Pain; Anesthesia
Keywords: postoperative pain; regional anesthesia; general anesthesia; gynecological laparoscopy
MeSH Terms: conditions — Pain, Postoperative | interventions — Midazolam; Sufentanil; Propofol; Rocuronium; Sevoflurane; Bupivacaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: general anesthesia (Other): Patients undergoing gynecological laparoscopic surgery under general anesthesia, using the following drugs: Midazolam, Propofol, Sufentanil, Rocuronium, Sevoflurane
  Interventions: Drug: Midazolam; Drug: Sufentanil; Drug: Propofol; Drug: Rocuronium; Drug: Sevoflurane
- Group B: regional anesthesia (Other): Patients undergoing gynecological laparoscopic surgery under regional anesthesia, using the following drugs: Sufentanil, Bupivacaine
  Interventions: Drug: Sufentanil; Drug: Bupivacaine

INTERVENTIONS:
Drug: Midazolam — Used for general anesthesia for gynecological laparoscopic procedures, together with Propofol, Sufentanil, Rocuronium, Sevoflurane
  Arms: Group A: general anesthesia
Drug: Sufentanil — Used for regional anesthesia (spinal or combined spinal-epidural anesthesia) for gynecological laparoscopic procedures together with Bupivacaine; and for general anesthesia for gynecological laparoscopic procedures, together with following drugs: Midazolam, Propofol, Rocuronium, Sevoflurane
Drug: Propofol — Used for general anesthesia for gynecological laparoscopic procedures, together with the following drugs: Midazolam, Sufentanil, Rocuronium, Sevoflurane
  Arms: Group A: general anesthesia
Drug: Rocuronium — Used for general anesthesia for gynecological laparoscopic procedures, together with the following drugs: Midazolam, Propofol, Sufentanil, Sevoflurane
  Arms: Group A: general anesthesia
Drug: Sevoflurane — Used for general anesthesia for gynecological laparoscopic procedures, together with the following drugs: Midazolam, Propofol, Sufentanil, Rocuronium
  Arms: Group A: general anesthesia
Drug: Bupivacaine — Used for regional anesthesia (spinal or combined spinal-epidural anesthesia) for gynecological laparoscopic procedures, together with Sufentanil
  Arms: Group B: regional anesthesia

SUMMARY:
Patients undergoing laparoscopic gynecological surgery will receive regional anesthesia or general anesthesia with endotracheal intubation. The investigators aim to evaluate the feasibility and safety of regional anesthesia for laparoscopic gynecological procedures.

DETAILED DESCRIPTION:
Commonly, laparoscopic gynecological procedures are performed under general anesthesia with endotracheal intubation.

The use of regional anesthesia in laparoscopy is reserved to patients declared unfit for general anesthesia because of severe comorbidities or it is applied in combination with general anesthesia to decrease postoperative pain.

Recently, growing literature evidence supports the use of regional anesthesia in patients undergoing laparoscopy.

The combination of minimally invasive surgery with regional anesthesia could increase the advantages of laparoscopic operations (less postoperative pain, shorter hospital stay, etc).

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing gynecological laparoscopic surgery;
* expected surgical time shorter than 90 minutes;
* informed consent to participate in the study.

Exclusion Criteria: none.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Feasibility and safety: Clavien-Dindo Classification (from Grade I to V) | From the surgery time, assessed up to 7 days after surgery
  Evaluation of feasibility and safety of regional anesthesia for gynecological laparoscopic surgery, considering complications using Clavien-Dindo Classification (from Grade I to V)

SECONDARY OUTCOMES:
Postoperative nausea or emesis. | 48 hours after surgery
  evaluation of the presence of postoperative nausea or emesis.
Days of hospitalization | From surgery to hospitalization discharge, assessed up to 7 days after surgery.
  Number of days of hospitalization after surgery.
Day of mobilization. | From surgery to day of first mobilization, assessed up to 7 days after surgery.
  Day of first mobilization after surgery.
Day of feeding. | From surgery to day of first feeding, assessed up to 7 days after surgery.
  Day of first feeding after surgery.
Day of canalization. | From surgery to day of first canalization, assessed up to 7 days after surgery.
  Day of first canalization after surgery.
Intraoperative pain: verbal numeric rating scale | Intraoperative: from skin incision to cutaneous suture.
  Intraoperative pain in patients submitted to regional anesthesia (Group B), using a verbal numeric rating scale, from 0 to 10, where 0 is no pain and 10 is the worse pain ever
Minimum respiratory rate | Intraoperative: from skin incision to cutaneous suture.
  Minimum respiratory rate during surgery.
End-Tidal PCO2 before pneumoperitoneum. | Intraoperative: from anesthesia to the beginning of pneumoperitoneum induction.
  End-Tidal PCO2 is measured by capnography.
End-Tidal PCO2 during pneumoperitoneum. | Intraoperative: pneumoperitoneum time expressed in minutes.
  End-Tidal PCO2 is measured by capnography.
Postoperative pain: numerical rating scale | 48 hours after surgery
  Evaluation of postoperative pain in patients undergoing general or regional anesthesia for gynecological laparoscopic surgery, measured with verbal numerical rating scale, from 0 to 10, where 0 is no pain and 10 is the worse pain ever

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Cardiothoracic and Vascular Anesthesia and Intensive Care, S. OrsolaMalpighi University Hospital, Bologna, BO
  - Gynecology and Physiopathology of Human Reproductive Unit, University of Bologna, S. Orsola-Malpighi Hospital, Bologna, BO